CLINICAL TRIAL: NCT02043613
Title: Effect of Physical Surroundings on Effects From Exercise as Treatment for Hip or Knee Pain: A Double-blind Randomized Controlled Clinical Trial
Brief Title: Context Effects in Exercise Therapy for Knee and/or Hip Pain
Acronym: CONEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: The Swedish Research Council (Other Government); The Danish Rheumatism Association (funding) (Unknown)
Responsible Party: Principal Investigator, Louise Fleng Sandal, MSc, Ph.d student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20130130
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Joint Pain; Knee Pain; Hip Pain; Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Joint pain; Context effects; Placebo effect; Exercise treatment
MeSH Terms: conditions — Arthralgia; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise in standard room (Active Comparator): Intervention: Exercise
  Patients exercise in standard physical surroundings. The room is marked by years of use. The room is placed in the basement, has artificial lighting, poor acoustics and bare concrete walls.
  Interventions: Other: Neuromuscular exercise
- Exercise in a contexually enhanced room (Experimental): Intervention: Exercise + contextually enhanced physical surroundings
  Patients exercise in a contextually enhanced room. The room has both artificial lighting and daylight, view of a recreational park, better acoustics, decorations among other factors, which may cause or enhance the context effect.
  Interventions: Other: Contextually enhanced physical surroundings of exercise; Other: Neuromuscular exercise
- Waiting list (No Intervention): Patients on waiting list are included, baseline tested and placed on a waiting-list for a 8 week period and tested at 8 weeks follow-up. The group is representative of the natural cause of disease.

INTERVENTIONS:
Other: Contextually enhanced physical surroundings of exercise — Different physical surroundings of exercise may affects the patients differently and consequently influence the effect of exercise. The exercise rooms are different from each other on parameters such as source of lighting, acoustics, materials and decorations.
  The differences with the physical surroundings of exercise is the primary intervention for this study.
  Arms: Exercise in a contexually enhanced room
Other: Neuromuscular exercise — The neuromuscular exercise program is the same across the two exercise groups. Consequently, this intervention is not the primary intervention of this study. The exercise program is based on the previously reported NEMEX program designed for patients with hip or knee osteoarthritis, originally published by Ageberg et al, 2010 in BMCMusculoskeletal Disorders.
  Arms: Exercise in a contexually enhanced room; Exercise in standard room

SUMMARY:
The study is designed to investigate the effect of physical surroundings on the effect of exercise therapy for knee and hip pain.

DETAILED DESCRIPTION:
Context effect have been shown to be influential in health-care settings, such as hospitals. This study investigates if context effects can be caused by the physical surroundings of exercise.

The study is designed as a double-blind randomized controlled clinical trial. Patients with knee and/or hip pain with a duration of a least 3 months are included in the trial and randomly assigned to 3 groups.

1. Exercise in pre-existing, standard room
2. Exercise in contextually enhanced room.
3. Waiting list.

The intervention consists markedly different between the two exercise rooms. The physical surroundings are described by factors such as acoustics, light source and intensity, decorations and air quality.

The exercise program applied is based on a previously investigated neuromuscular exercise program, NEMEX. The same program is performed in both exercise rooms. Consequently, only the physical surroundings differ between intervention groups.

Patients' "global perceived effect" is used as the primary outcome assessed at 8 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35 years or older
* Self-report of knee and/or hip pain within the last 3 months.
* Willing and able to attend exercise therapy at the University of Southern Denmark, Odense M twice weekly.

Exclusion Criteria:

* Co-morbidities or contraindication prohibiting to participation in exercise therapy.
* Unable to fill-out questionnaires, or to speak, read or understand Danish.
* Already participating in exercise therapy*, having had surgery to the hip/knee within the last 3 months or on waiting list for joint surgery within the coming 6 months. (*defined as supervised exercise program by physiotherapist, systematic strength training etc. with duration of 6 weeks or more)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Patients' Global Perceived Effect | 8 weeks
  Patients indicate their perception of the global effect of the intervention on a 7 point likert scale ranging from "substantially worse" to "no change" to "substantially improved". The scale is balanced around the 'no change' response with 3 steps in each direction, respectively deterioration or improvement.

SECONDARY OUTCOMES:
Change from baseline in KOOS (The Knee injury and Osteoarthritis Outcome Score) or HOOS (The Hip Dysfunction and Osteoarthritis Score), respectively | Baseline, 4 weeks, 8 weeks
Change from baseline in The 36-item Short-Form Health Survey (SF-36) | Baseline, 4 weeks, 8 weeks
Change from baseline in Arthritis Self-Efficacy Scale | baseline, 4 weeks, 8 weeks.
  A modified version of the Arthritis Self-Efficacy Scale consisting of 11 items scoring patient reported self-efficacy
Patient satisfaction with physical surroundings | 8 weeks
  Patients are asked to indicate their level of satisfaction with different elements of the physical surroundings.

OTHER OUTCOMES:
Change from baseline in functional test: Single limb mini squat | Baseline, 8 weeks
Change from baseline in functional test: Maximal number of knee bendings pr. 30 sec. | baseline, 8 weeks
Change from baseline in functional test: Number of chair stands per. 30 sec. | baseline, 8 weeks
Change from baseline in functional test: Timed 40 m walking test | baseline, 8 weeks
Change from baseline in functional test: One leg hop for distance | Baseline, 8 weeks,
Change from baseline in muscle strength, MVC knee extension | baseline, 8 weeks
change from baseline in muscle strength, MVC, hip abduction | baseline, 8 weeks
Change from baseline in aerobic capacity measured by a submaximal bicycle test by Aastrand & Saltin | Baseline, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louise F. Sandal, MSc, Principal Investigator — Research Unit of Musculoskeletal Function and Physiotherapy
Locations (1):
- Research Unit of Musculoskeletal Function and Physiotherapy, Department of Sports Science and Clinical Biomechanics, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Derived] Sandal LF, Thorlund JB, Moore AJ, Ulrich RS, Dieppe PA, Roos EM. Room for improvement: a randomised controlled trial with nested qualitative interviews on space, place and treatment delivery. Br J Sports Med. 2019 Mar;53(6):359-367. doi: 10.1136/bjsports-2016-097448. Epub 2017 Aug 2. PMID 28768617
- [Derived] Sandal LF, Thorlund JB, Ulrich RS, Dieppe PA, Roos EM. Exploring the effect of space and place on response to exercise therapy for knee and hip pain--a protocol for a double-blind randomised controlled clinical trial: the CONEX trial. BMJ Open. 2015 Mar 27;5(3):e007701. doi: 10.1136/bmjopen-2015-007701. PMID 25818278